CLINICAL TRIAL: NCT02324959
Title: Evaluation of Acupuncture and Attention Training Effects on Patients After Stroke: a Study Protocol of an International Multicentre Study Using a Randomized Single Blinded Three-group Design
Brief Title: Acupuncture and Computer-based Training to Improve Attention Deficits in Patients After Stroke
Acronym: ACoTrain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian University of Traditional Chinese Medicine (Other)
Collaborators: Reha Rheinfelden (Other); m&i-Fachklinik Herzogenaurach (Unknown)
Responsible Party: Principal Investigator, Shanli Yang, Dr., Fujian University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 651
Record Dates: First submitted 2014-12-08; First posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acupuncture (Active Comparator): Needling of affected meridian groups in line with Traditional Chinese Medicine procedures (Baihui and Shenting).
  Interventions: Device: Acupuncture
- Computer-based (Active Comparator): Computer-based attention training (RehaCom).
  Interventions: Device: RehaCom
- ACoTrain (Experimental): A combination of computer-based attention training with acupuncture.
  Interventions: Device: RehaCom; Device: Acupuncture

INTERVENTIONS:
Device: RehaCom — The computer-based neurorehabilitation program is intended for patients with acquired cognitive deficits after brain damage, e.g. after stroke. The RehaCom software has five different therapeutic groups aimed at restoration of attention, memory, executive functions, and visual field, respectively. Each group has one to four different modules to choose from for each therapy session. Only attention will be trained in this study.
  Other Names: computer-based attention training
  Arms: ACoTrain; Computer-based
Device: Acupuncture — The affected meridian group is treated by needling on Baihui (GV20|DU20) and Shenting (GV24|DU24) - both acupoints of the Governor Vessel. Baihui is 5 cun (1cun=3.33 cm) superior to the anterior hairline on the anterior median line (midpoint of the connecting line between the auricular apices).
  Arms: ACoTrain; Acupuncture

SUMMARY:
The purpose of this study is to determine whether acupuncture and computer-based attention training can be combined for more effective post-stroke attentional deficits.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to inpatient stroke rehabilitation within six months after first-ever stroke
* Mild cognitive impairments (attention performance TAP > 1 standard deviation below mean age-matched norm in at least one subtest).
* Conscious, stable physical condition and signed informed consent of patient.

Exclusion Criteria:

* Severe visual and/or hearing problems
* Inability to follow instructions (MoCA)
* Disorders of speech and instruction comprehension (tested with a modified token-test)
* Severe visual and/or hearing problems
* Pre-existing mental disorders - Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-11 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in attention performance at 4 weeks (Test Battery for Attention Performance (TAP)) | Pretest (day 1), Posttest (4 weeks)

SECONDARY OUTCOMES:
Change from Baseline in time needed for Trail Making Test (TMT A/-B) at four weeks. | Pretest (day 1), Posttest (4 weeks)
Change from Baseline in number of errors for the Test des Deux Barrage (T2B) at four weeks. | Pretest (day 1), Posttest (4 weeks)
Change from Baseline in number of omissions for the Test des Deux Barrage (T2B) at four weeks. | Pretest (day 1), Posttest (4 weeks)
National Institute of Health Stroke Scale (NIH-SS) | Pretest (day 1)
Change from baseline in total score of Extended Barthel Index (EBI) at four weeks. | Pretest (day 1), Posttest (4 weeks)
Change from baseline score of EuroQol quality of life questionnaire (EQ-5D 3L) at four weeks. | Pretest (day 1), Posttest (4 weeks)

CONTACTS AND LOCATIONS:
Locations (3):
- Fujian University of Traditional Chinese Medicine, Fuzhou, Fujian, China
- m&i Fachklinik Herzogenaurach, Herzogenaurach, Bavaria, Germany
- Reha Rheinfelden, Rheinfelden, Canton of Aargau, Switzerland

REFERENCES:
- [Derived] Huang J, McCaskey MA, Yang S, Ye H, Tao J, Jiang C, Schuster-Amft C, Balzer C, Ettlin T, Schupp W, Kulke H, Chen L. Effects of acupuncture and computer-assisted cognitive training for post-stroke attention deficits: study protocol for a randomized controlled trial. Trials. 2015 Dec 2;16:546. doi: 10.1186/s13063-015-1054-x. PMID 26631161